CLINICAL TRIAL: NCT00005570
Title: An Epidemiological Study of Subjects With Immune Thrombocytopenic Purpura to Evaluate the Relationship Between Platelet Counts, Endogenous Thrombopoietin Levels, Endogenous Anti-Thrombopoietin Antibodies, and Selected Autoimmune Markers
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000120; 00-H-0120
Record Dates: First submitted 2000-04-22; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-04

CONDITIONS: Purpura, Thrombocytopenic, Idiopathic; Immune Thrombocytopenic Purpura
Keywords: Bleeding; Cytokines; Immune Response; Pharmacogenomic; Serum Antibodies; ITP; Immune Thrombocytopenia Purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Hemorrhage

SUMMARY:
This study involves the collection of blood samples from patients with immune thrombocytopenic purpura (ITP) to evaluate the relationship between platelet counts, blood levels of a hormone called thrombopoietin that controls platelet production by the bone marrow, and blood levels of antibodies against thrombopoietin that could interfere with the action of this hormone. Blood samples will also be stored if separately agreed to by the patient for analysis of genes that might affect platelet production. At a single outpatient clinic visit, patients will have a medical history taken, and blood samples drawn for testing. Results from this study may help further understand the control of platelet production in patients with ITP, and suggest new therapeutic approaches.

DETAILED DESCRIPTION:
This study involves the collection of blood samples from patients with immune thrombocytopenic purpura (ITP) to evaluate the relationship between platelet counts, blood levels of a hormone called thrombopoietin that controls platelet production by the bone marrow, and blood levels of antibodies against thrombopoietin that could interfere with the action of this hormone. Blood samples will also be stored if separately agreed to by the patient for analysis of genes that might affect platelet production. At a single outpatient clinic visit, patients will have a medical history taken, and blood samples drawn for testing. Results from this study may help further understand the control of platelet production in patients with ITP, and suggest new therapeutic approaches.

ELIGIBILITY:
Diagnosis of ITP, based on the history, physical examination, complete blood count, and examination of the peripheral smear, which should exclude other causes of thrombocytopenia. These criteria for ITP are based on the American Society of Hematology practice guideline for ITP.

Subjects 5 years of age or older.

Before the study specific procedure, the subject or legally acceptable representative must give written informed consent(s) for participation in the study.

No subjects with documented history of Human Immunodeficiency Virus (HIV) or Hepatitis.

No subjects with known underlying causes of thrombocytopenia such as lupus erythematosus, autoimmune thyroid disorders, drug-induced thrombocytopenia, bone marrow disorders, and liver disease.

No psychiatric or addictive disorders that compromise the subject's ability to give truly informed consent for participation in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2000-04; Study Completion 2000-07

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Kelton JG, Gibbons S. Autoimmune platelet destruction: idiopathic thrombocytopenic purpura. Semin Thromb Hemost. 1982 Apr;8(2):83-104. doi: 10.1055/s-2007-1005045. No abstract available. PMID 6210960